CLINICAL TRIAL: NCT01232439
Title: Assessment of Brain Kappa Opioid Receptor Occupancy After Single Oral Doses of LY2456302 as Measured by PET With Radioligand LY2879788 in Healthy Subjects
Brief Title: A Study of Brain Receptor Occupancy in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12511; I2Z-MC-LAFC (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-20; First posted 2010-11-02 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Aticaprant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- opioid receptor kappa antagonist (Experimental)
  Interventions: Drug: opioid receptor kappa antagonist

INTERVENTIONS:
Drug: opioid receptor kappa antagonist — Starting dose of 2 mg, administered orally, once.
  The potential dose range for this study is 0.2 mg to 30 mg
  Other Names: LY2456302

SUMMARY:
To measure the occupancy of brain kappa opioid receptors after single oral doses of LY2456302.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Have clinical laboratory tests within normal reference ranges
* Have arterial and venous access sufficient to allow blood sampling

Exclusion Criteria:

* Currently enrolled in, or discontinued within the last 30 days from a clinical trial
* History of severe allergies or multiple adverse drug reactions
* Have an abnormal ECG at screening visit
* Have abnormal sitting blood pressure
* Have an increased risk of seizures
* Current suicidal ideation
* Positive test for HIV, hepatitis C, or hepatitis B
* Women who are breast feeding
* Smoke more than 10 cigarettes per day, or equivalent
* Drink more than 5 cups of coffee per day, or equivalent
* Have a history of head injury
* Unable to undergo a MRI
* Suffer from claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in brain kappa opioid receptor occupancy (RO) by positron emission tomography (PET) | Baseline, after single dose of study drug

SECONDARY OUTCOMES:
Pharmacokinetics, area under the curve (AUC) | Days 1 and 2
Number of participants with clinically significant effects | Baseline to study completion
Pharmacokinetics, concentration maximum (Cmax) | Days 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut, United States